CLINICAL TRIAL: NCT00989118
Title: Randomized Study on Endometrioma Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Model: Parallel
Other Study IDs: endometriomatreatment
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2009-10-02 (Estimated); Status verified 2009-10

CONDITIONS: Ovarian Endometrioma
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laser treatment (Experimental)
  Interventions: Procedure: Laser treatment of ovarian endometrioma
- Endometrioma cystectomy (Active Comparator)
  Interventions: Procedure: Laser treatment of ovarian endometrioma

INTERVENTIONS:
Procedure: Laser treatment of ovarian endometrioma — Laser vaporization of ovarian endometrioma

SUMMARY:
This is a randomised study comparing the effect of two laparoscopic techniques for treatment of ovarian endometriomas on recurrence rate and ovarian reserve.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 40 years
* uni or bilateral symptomatic endometriotic cysts with a minimum diameter of 30 millimetres
* no counter-indication for the use of GnRH analogues

Exclusion Criteria:

* previous pelvic surgeries
* history of cancer
* suspected malignancy
* presurgical suspicion or evidence of deep endometriosis
* presurgical suspicion or evidence of premature ovarian failure
* use of oestrogen suppressive drugs in the preceding 6 months

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2000-05; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Carmona F, Martinez-Zamora MA, Rabanal A, Martinez-Roman S, Balasch J. Ovarian cystectomy versus laser vaporization in the treatment of ovarian endometriomas: a randomized clinical trial with a five-year follow-up. Fertil Steril. 2011 Jul;96(1):251-4. doi: 10.1016/j.fertnstert.2011.04.068. Epub 2011 May 14. PMID 21575941